CLINICAL TRIAL: NCT03671109
Title: Evaluation of the Safety and Efficacy of Dihydroartemisinin-piperaquine for Intermittent Preventive Treatment of Malaria in HIV-infected Pregnant Women
Brief Title: Improving Maternal heAlth by Reducing Malaria in African HIV Women
Acronym: MAMAH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: Medicines for Malaria Venture (Other); Universität Tübingen (Other); Centre de Recherche Médicale de Lambaréné (Other); Medical University of Vienna (Other); Bernhard Nocht Institute for Tropical Medicine (Other Government); Centro de Investigação em Saúde de Manhiça (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EDCTP- RIA2016MC-1613
Record Dates: First submitted 2018-09-06; First posted 2018-09-14 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Malaria; HIV/AIDS; Pregnancy Related
Keywords: Malaria; Dihydroartemisinin-piperaquine; HIV; Pregnancy; Treatment; Prevention
MeSH Terms: conditions — Malaria; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Superiority clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPTp-DHA-PPQ (Experimental): Monthly IPTp-DHA-PPQ over three days plus daily ARVs and cotrimoxazole prophylaxis
  Interventions: Drug: Dihydroartemisinin-piperaquine (DHA-PPQ)
- IPTp-Placebo (Placebo Comparator): Monthly IPTp-placebo over three days plus daily ARVs and cotrimoxazole prophylaxis
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine (DHA-PPQ) — Following physical examination, recruited women with more than 13 weeks of gestational age will receive IPTp-DHA-PPQ under supervision
  Arms: IPTp-DHA-PPQ
Drug: Placebo Oral Tablet — Following physical examination, recruited women with more than 13 weeks of gestational age will receive IPTp-Placebo under supervision
  Arms: IPTp-Placebo

SUMMARY:
Trial to evaluate the safety and efficacy of DHA-PPQ for Intermittent Preventive Treatment (IPTp) in HIV-infected pregnant women receiving cotrimoxazole prophylaxis (CTXp) and antiretroviral (ARV) drugs and using long lasting insecticide treated nets will be conducted in Mozambique and Gabon where malaria and HIV infection are moderate to highly prevalent. In addition, the possibility for a PK interaction between DHA-PPQ and ARV drugs will be assessed in a sub-sample of participants. Women will receive ARV therapy according to national guidelines and their infants will be followed until one year of age to evaluate the impact of DHA-PPQ on MTCT-HIV.

DETAILED DESCRIPTION:
Background

Intermittent preventive treatment in pregnancy (IPTp) with sulphadoxine-pyrimethamine (SP) is recommended for malaria prevention in HIV-uninfected women but it is contraindicated in those HIV-infected on cotrimoxazole prophylaxis (CTXp) due to potential adverse effects. A recent trial showed that an effective antimalarial added to CTXp and long-lasting insecticide treated nets (LLITNs) in HIV-infected pregnant women improves malaria prevention and maternal health. However, the antimalarial used -mefloquine- was not well tolerated and it was associated with an increase in HIV viral load at delivery and a two-fold increased risk of MTCT-HIV. These findings highlight the need to find alternative drugs with better tolerability and safety profile to prevent malaria in this vulnerable group and to further study the pharmacological interactions between antimalarials and antiretrovirals (ARVs).

Dihydroartemisinin-piperaquine (DHA-PPQ), because of its long half-life and good tolerability has been shown to improve antimalarial protection in HIV-uninfected pregnant women, constituting the most promising candidate for IPTp in HIV-infected pregnant women. However, there is limited information on the pharmacokinetics of DHA-PPQ with concomitant use of ARV drugs and CTX, particularly in pregnant women.

Objectives

1. To evaluate the safety, tolerability and efficacy of DHA-PPQ as IPTp for malaria prevention in HIV-infected pregnant women receiving daily CTXp and ARV drugs
2. To assess the effect of DHA-PPQ as IPTp on mother to child transmission of HIV
3. To study the effects of DHA-PPQ on the pharmacokinetics of clinically relevant doses of ARV drugs used for prevention of MTCT and treatment of HIV infection
4. To evaluate the effectiveness of CTXp in clearing malaria parasites in HIV-infected pregnant women

Methods

The trial has been designed as a randomized double blind placebo-controlled superiority trial to evaluate the safety and efficacy of DHA-PPQ as IPTp in HIV-infected pregnant women taking daily CTXp and ARV drugs. The trial sites are located in Central and South Eastern sub-Saharan Africa (Gabon and Mozambique), where HIV prevalence among pregnant women ranges from 6 to 29%.

Based on previous estimations at the study sites and assuming a prevalence of peripheral parasitaemia at delivery of 7.5% with CTXp, it is estimated that 298 women per arm will be required to detect with 80% power a significant (p<0.05) decrease of 5% or more in the prevalence of peripheral parasitaemia in the CTXp+IPTp-DHA-PPQ group. In order to allow for 10% losses to follow up, it is calculated that 332 women/study arm will need to be recruited (total n=664). Furthermore, assuming a 5% MTCT-HIV in the control group, this sample size will have an 80% power to detect at the 5% level of significance, 2.2 times difference in the risk of MTCT-HIV.

The trial will have two study arms; HIV-infected pregnant women participating in the trial will be randomized to receive either:

1. Monthly doses of IPTp-DHA-PPQ over three days plus daily ARVs and cotrimoxazole prophylaxis
2. Monthly doses of IPTp-placebo over three days plus daily ARVs and cotrimoxazole prophylaxis

Women will receive ARV therapy according to national guidelines and their infants will be followed until one year of age to evaluate the impact of DHA-PPQ on MTCT-HIV.

Participants will be asked to visit the ANC monthly and to deliver at the study health facilities. Adherence to CTX prophylaxis and ARV therapy, as well as use of the LLITNs use will be assessed monthly at the scheduled antenatal care (ANC) clinic visits.

Pharmacokinetic (PK) sub-study The possibility for a PK interaction between DHA-PPQ and ARV drugs will be assessed in a sub-sample of participants (n=200).

ELIGIBILITY:
Inclusion Criteria:

* Permanent resident in the study area
* Gestational age at the first antenatal visit ≤ 28 weeks
* HIV seropositive status
* Agreement to deliver in the study site's maternity(ies) wards

Exclusion Criteria:

* Residence outside the study area or planning to move out in the following 10 months from enrolment
* Gestational age at the first antenatal visit > 28 weeks of pregnancy
* Known history of allergy to CTX
* Known history of allergy or contraindications to DHA-PPQ
* Participating in other intervention studies

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Maternal parasitaemia at delivery | Delivery
  Presence of Plasmodium falciparum (P. falciparum) asexual parasites of any density in peripheral blood (determined by microscopy)

SECONDARY OUTCOMES:
Incidence of clinical malaria | On average six months follow up during pregnancy
Incidence of all-cause admissions | On average six months follow up during pregnancy
Incidence of all-cause outpatient attendances | On average six months follow up during pregnancy
Frequency and severity of adverse events | On average six months follow up during pregnancy
Mean haemoglobin concentration | At delivery
Prevalence of submicroscopic P. falciparum peripheral parasitaemia | At delivery
Prevalence of anaemia (Hb<11 g/dL) | At delivery
Prevalence of severe anaemia (Hb<7 g/dL) | At delivery
Mean CD4+ T cell counts levels | At delivery
Proportion of women with detectable HIV viral load | At delivery
Prevalence of placental P. falciparum infection | At delivery
Prevalence of P. falciparum peripheral parasitaemia at the post-partum visit | On average 42 days after end of pregnancy (post-partum visit)
Maternal mortality rate | On average six months follow up during pregnancy and 42 days after end of pregnancy (post-partum visit)
Prevalence of P. falciparum parasitaemia in cord blood | At birth
Prevalence of neonatal anaemia | Neonatal period ( in first 28 days of life)
Mean birth weight | At birth
Prevalence of low birth weight (<2500 g) | At birth
Mean gestational age at birth | At birth
Prevalence of prematurity | At birth
Prevalence of embryo and foetal losses | On average six months follow up during pregnancy
Prevalence of small for gestational age | At birth
Frequency of congenital malformations | At birth
Incidence of clinical malaria | During first year of life
Neonatal mortality rate | During neonatal period (during first 28 days of life)
Frequency of mother to child transmission of HIV at one and at 12 months of age | During first year of life
Infant mortality rate | During first year of life
Composite malaria outcome: proportion of participants with malaria infection diagnosed | From enrolment until one month after end of pregnancy (on average seven months of study follow up of women, depending on gestational age at inclusion)
  Any malaria confirmed infection during follow up, delivery and post-partum period (blood smear, malaria PCR, placental infection)
Composite maternal malaria and anemia: proportion of particiapnts diganosed either with malaria or anemia | At delivery
Composite adverse pregnancy outcome | Birth
  LBW, miscarriage, stillbirth, prematurity

CONTACTS AND LOCATIONS:
Overall Officials: Clara Menendez, MD, PhD, Study Director — Barcelona Institute for Global Health
Locations (2):
- Centre de Recherches Médicales de Lambaréné (CERMEL), Lambaréné, Gabon
- Centro de Investigação em Saúde de Manhiça (CISM), Manhiça, Mozambique

IPD SHARING:
Plan to Share IPD: Yes
The main findings of the clinical trial will be submitted for publication in a peer reviewed journal within 12 months of study completion through an open access mechanism, or otherwise made available publicly in compliance with H2020 open access requirements.
  Primary project raw data will be published in the project website. This approach is taken to protect in particular the interests of the endemic country researchers and institutions and in acknowledgment of the primary research oversight by endemic country ethics review boards. At no stage will data containing personal information of research participants be released.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Project metadata will be made available in formal reports to key stakeholders as soon as possible and to the wider public within 12 months after the end of the project. The announcement of the availability of the project metadata will be posted in the project website.
Access Criteria: Open Access

REFERENCES:
- [Result] Gonzalez R, Nhampossa T, Mombo-Ngoma G, Mischlinger J, Esen M, Tchouatieu AM, Mendes A, Figueroa-Romero A, Zoleko-Manego R, Lell B, Lagler H, Stoeger L, Dimessa LB, El Gaaloul M, Sanz S, Mendez S, Piqueras M, Sevene E, Ramharter M, Saute F, Menendez C; MAMAH study group. Safety and efficacy of dihydroartemisinin-piperaquine for intermittent preventive treatment of malaria in pregnant women with HIV from Gabon and Mozambique: a randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2024 May;24(5):476-487. doi: 10.1016/S1473-3099(23)00738-7. Epub 2024 Jan 12. PMID 38224706
- [Result] Gonzalez R, Nhampossa T, Mombo-Ngoma G, Mischlinger J, Esen M, Tchouatieu AM, Pons-Duran C, Dimessa LB, Lell B, Lagler H, Garcia-Otero L, Zoleko Manego R, El Gaaloul M, Sanz S, Piqueras M, Sevene E, Ramharter M, Saute F, Menendez C. Evaluation of the safety and efficacy of dihydroartemisinin-piperaquine for intermittent preventive treatment of malaria in HIV-infected pregnant women: protocol of a multicentre, two-arm, randomised, placebo-controlled, superiority clinical trial (MAMAH project). BMJ Open. 2021 Nov 23;11(11):e053197. doi: 10.1136/bmjopen-2021-053197. PMID 34815285
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693
- See also: Project webpage — http://www.mamahproject.net/